CLINICAL TRIAL: NCT02956395
Title: Protocol for Regional Implementation of Community-based Collaborative Management of Complex Chronic Patients (CCP)
Brief Title: Implementation of Community-based Collaborative Management of Complex Chronic Patients
Acronym: Nextcare_CCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Badalona Serveis Assistencials (Other); Institut de Recerca Biomèdica de Lleida (Other)
Responsible Party: Principal Investigator, Carme Hernandez, Director Integrated Care Unit, Hospital Clinic of Barcelona
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Nextcare_CCP
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Chronic Disease; Integrated Care; Telemedicine
Keywords: adaptive case management approach; Transitional Care; multimorbidity
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated care group (Active Comparator): Integrated care intervention is implemented by a multidisciplinary team from the hospital and from the Primary Care in three healthcare sectors: Barcelona-Esquerra, Lleida and Badalona.
  Interventions: Other: Integrated care intervention
- Conventional care group (No Intervention): Patients assigned to the control group will be from other healthcare sectors in Catalonia with similar characteristics.

INTERVENTIONS:
Other: Integrated care intervention — Integrated care intervention is implemented by a multidisciplinary team from the hospital and from the Primary Care.
  The intervention after hospital discharge a) Phone call at 24 hours; b) Home visit at 72 hours after discharge by one member of the transitional care team, if is needed; During this visit, the therapeutic plan for each patient will be customized to their individual frailty factors and shared with the primary care team. Reinforcement of the logistics for treatment of co-morbidities and social support will be done accordingly; c) Accessibility to the point of care available 24 hours/day ; d) Accessibility to the individualized PHF, as self-management tool ; d) appointment at 1m after discharge and after 12 m
  Arms: Integrated care group

SUMMARY:
Background/Aims: Large scale adoption of integrated care for chronic patients constitutes a key milestone to accelerate adaptation of current healthcare systems to the evolving needs triggered by population ageing and high prevalence of chronic conditions. Lessons learnt from deployment experiences are being disseminated as "good practices". But, there is need for further assessment of implementation strategies in real world scenarios. Moreover, progresses achieved in disease-oriented integrated care cannot be automatically transferred to management of complex chronic patients (CCP). The protocol addresses five aims: 1) implementation of two integrated care interventions using a collaborative and adaptive case management (ACM) approach (i) Community-based management of CCP; and, ii) Integrated care for patients under long-term oxygen therapy (LTOT)); 2) adoption of information and communication technologies (ICT) required to support collaborative ACM; 3) to evaluate the impact of enhanced clinical health risk assessment and stratification; 5) to generate a roadmap for regional adoption of the CCP program.

Methods/Design: the CCP program will be deployed in three healthcare sector of Barcelona-Esquerra (AISBE) (520 k citizens) and in two other areas of Catalonia: Badalona Serveis Assistencials (BSA) (420 k citizens) and Lleida (366 k citizens) following Plan-Do-Study-Act iterative cycles, using the Model for Assessment of Telemedicine for evaluation purposes. The study also addresses the steps for scale-up of integrated care in the entire Catalan region (7.5 M citizens). Observational studies with matched controls have been planned for both Community-based management of CCP (n=3.000) and for Integrated care for patients under LTOT (n=500). Moreover, clustered randomized controlled trials (RCT) are planned on top of the observational studies to test specific questions (i.e. performance of the ICT platform providing ACM functionalities). Main components of CCP program are: a) patient stratification; b) comprehensive assessment strategies; c) ICT supported adaptive Case management; d) Roadmap for regional adoption.

Hypothesis: the CCP program will generate guidelines for large scale deployment of the CCP program, including transferability analysis, facilitating adoption of integrated care services for management of multi-morbidity.

DETAILED DESCRIPTION:
Rationale & hypothesis - Both, management of multi-morbidity and efficient collaboration between specialized care and community-based services are unmet needs that can be overcome by implementation of structured, but flexible, service workflows. That is, an ACM approach, as well as appropriate patient health risks assessment and stratification.

The service workflow has two sequential phases with specific target outcomes for each of them: i) Short-term (30 and 90 days after hospital discharge) prevention of hospital-related events after hospital discharge; and ii) Intervention aiming at long-term enhanced CCP management.

Objectives - To assess the impact of ICT-supported ACM on: i) reduction of early hospital-related events including hospital re-admissions, visits to emergency department and mortality; and, ii) Health value generation of the long-term intervention, defined as target outcomes achieved relative to their costs.Detailed outcomes include the eleven indicators recommended by the Spanish Health System covering the following dimensions: i) Characteristics of the study groups and health status (i.e, Users attended in primary care and, Health-related quality of life of patients and caregivers); ii) Intermediate outcomes (Emergency Department visits; General Practitioner visits; Cumulative days per year admitted in hospital; Poli-medication; Potentially avoidable hospitalizations; Hospital readmissions; Needs for social support); iii) Empowerment (Unhealthy life styles); and, iv) Structure (Access to ICT-supported integrated care). Moreover, through the program lifespan progresses consolidated by the International Consortium for Health Outcomes Measurement (ICHOM) will be incorporated.

Study design - The large-scale deployment will be evaluated as an observational study with a matched control group. Assessment will be done by an independent team. The number of patients to be included in the implementation study is approximately one-thousand individuals per year, including both conventional hospitalization and home hospitalization as recruitment sources.

Intervention - The general structure of the service workflow for the intervention group is as follows:

Case identification. Identification of candidates for inclusion into the program following the pre-defined inclusion/exclusion Case evaluation. During hospital admission or home hospitalization. A holistic characterization should be performed covering a threefold aim: i) Comprehensive assessment of each individual's need for health and social support; ii) Individualized pharmacological and non-pharmacological treatment, including adherence and self-management interventions needs; iii) Identification of short and long-term clinical requirements; and, iv) Assessment of barriers that may limit fulfilment of the program.

Personalized work plan definition - Personalized action plan based on case evaluation.

Work plan execution, follow-up and event handling with the support provided by information and communication technologies (ICT) that facilitate the program follow up and the handling of unexpected events by: i) fostering patient empowerment for self-management; ii) enhance patient adherence to the program; iii) facilitating remote supervision; and, iv) allowing patient monitoring.

Discharge - At the end of the program evaluation.Eventually, it can be moved to other types of integrated care services depending upon his/her needs.

The intervention is implemented by a multidisciplinary team from the hospital and from the Primary Care, of advanced-practice nurses, physicians, physiotherapists, community nurses, social workers having a general practitioner as a reference.

The collaboration between specialized care and primary care is guided by the reform of specialized care in the healthcare sectors initiated in 2006. Both teams share ICT-supported tools.

The intervention during hospital admission includes four key features: 1) A comprehensive assessment of the patient at entry; 2) A two-hour educational program administered at entry by a nurse followed by distribution of patient-specific support material.

Intervention after hospital discharge a) Phone call at 24 hours; b) Home visit at 72 hours after discharge. Accessibility to the point of care available 24 hours/day; PHF, as self-management tool and appointment at 1m after discharge.

After the transitional phase, the advanced-practice nurses perform regular training sessions to the community-based care teams, facilitate high accessibility to specialized care as needed and support functionalities of the PHF for the patients admitted into the program.

The number of home care visits, as well as access to specialized care, during the follow-up 12 month period is individually tailored, and dynamically adapted, to patient needs. Moreover, planned visits by specialized professionals can be scheduled through the day hospital or home visits if this was deemed necessary by primary care teams.

ICT- Support - The three main actors, namely: i) the healthcare professionals with access to an adaptive case management system for work plan prescription, follow-up, coaching, and care-coordination across healthcare tiers; ii) the adaptive case management system supporting execution of the patient work plan and providing a bridge of interoperability and collaborative tools among the patient (through the PHF), the case manager and the electronic medical record; and, iii) the patient, with access to the PHF wherein she/he can answer questionnaires, perform monitoring through mHealth apps, and have access to a follow-up reports and tailored educational information.

Control group - Patients assigned to usual care will follow conventional treatment, being managed by their physician without support by the multidisciplinary team, as described above for the intervention group.

Clinical assessment - Evaluation will be done by an independent team at baseline and after the 12-month follow-up. The questionnaires are those used by the integrated care team with additions designed to capture patient empowerment characteristics: mental status, activities of daily living, anxiety and depression, health-related quality of life; acute episodes requiring emergency department consultations and/or hospital admissions within the healthcare sector will be assessed using shared registries from the public health system. Moreover, core outcomes, will be assessed from public registries.

Data analysis- A sample size of 200 patients per group was necessary to recognize statistically significant effects of the intervention. The estimated number of patients identified during the screening process (one-thousand per year) is markedly higher than minimum required, thus ensuring enough statistical power.

Results will be expressed as mean and standard deviation (SD), or as number and percentages, in the corresponding categories. Comparisons between the two study groups on admission and at 12 months will be performed using unpaired Student t-test for continuous variables, if variables to be compared have two categories; and, chi-square tests for non-continuous variables. Changes within each group were assessed by paired analysis (for example using paired t test). The effects of the intervention on mortality and time to admission will be analyzed respectively using multivariate logistic and Cox regression models, adjusted for baseline differences between groups. We will build saturated models introducing all of the covariates which result statistically significant during bivariate assessment. After this, we will build parsimonious models by excluding, one to one, all of the variables not significant according to the Wald test p-value. Finally, we will decide the final model, comparing the saturated with the parsimonious models, according to the likelihood ratio test.Statistical significance is set at a p value less than 0.05. Analyses will be done with SPSS release 20.

Additionally, qualitative assessment of technology will be done using standard questionnaires and through focus groups.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients and LACE index ≥7.

Exclusion Criteria:

Severe psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Reduction of early hospital-related events after hospital discharge | 30 and 90 days and 12 months
  Hospital re-admissions

CONTACTS AND LOCATIONS:
Overall Officials: Carme Hernandez, RN, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona. Integrated Care Unit, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vela E, Tenyi A, Cano I, Monterde D, Cleries M, Garcia-Altes A, Hernandez C, Escarrabill J, Roca J. Population-based analysis of patients with COPD in Catalonia: a cohort study with implications for clinical management. BMJ Open. 2018 Mar 6;8(3):e017283. doi: 10.1136/bmjopen-2017-017283. PMID 29511004